CLINICAL TRIAL: NCT03681093
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Placebo-controlled Study of Fevipiprant Once Daily Plus Standard-of-care (SoC) for Assessment of the Efficacy in Reduction of Nasal Polyp Size in Patients With Nasal Polyposis and Concomitant Asthma.
Brief Title: Study of Efficacy of Fevipiprant in Patients With Nasal Polyposis and Asthma
Acronym: THUNDER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAW039A2322; 2018-002073-22 (EudraCT Number)
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Nasal Polyps
Keywords: Nasal Polyposis; Asthma; Nasal polyp score (NPS); Nasal congestion score (NCS); Bronchial Diseases; Lung Diseases; Nose Diseases; Respiratory Hypersensitivity; Fevipiprant; QAW039
MeSH Terms: conditions — Nasal Polyps; Asthma; Bronchial Diseases; Lung Diseases; Nose Diseases; Respiratory Hypersensitivity | interventions — fevipiprant

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind, double dummy study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fevipiprant 150 mg (Experimental): Fevipiprant (QAW039) 150 mg once daily orally
  Interventions: Drug: Fevipiprant 150 mg
- Fevipiprant 450 mg (Experimental): Fevipiprant (QAW039) 450 mg once daily orally
  Interventions: Drug: Fevipiprant 450 mg
- Placebo (Placebo Comparator): Placebo once daily orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fevipiprant 150 mg — Fevipiprant (QAW039) 150 mg once daily administered orally as tablet
  Arms: Fevipiprant 150 mg
Drug: Fevipiprant 450 mg — Fevipiprant (QAW039) 450 mg once daily administered orally as tablet
  Arms: Fevipiprant 450 mg
Drug: Placebo — Placebo once daily administered orally as tablet
  Arms: Placebo

SUMMARY:
A Phase 3b Proof-of-Concept study to evaluate the ability of fevipiprant 150 mg and 450 mg, compared with placebo, as add-on to nasal spray standard-of-care (SoC), in reducing endoscopic nasal polyp score in adult (≥ 18 years) patients with nasal polyposis and concomitant asthma.

DETAILED DESCRIPTION:
This was a Phase 3b, Proof-of-concept study with a randomized, multicenter, double-blind, placebo-controlled, parallel-group study design to determine the ability of fevipiprant plus standard of care (SoC) compared to placebo plus SoC to reduce the size of nasal polyps. The study enrolled adult male and female patients diagnosed with nasal polyposis with a nasal polyp score assessed by nasal endoscopy ≥ 4 at baseline with a minimum score of 2 in each nostril and a concomitant diagnosis of asthma. Patients who meet the inclusion/exclusion criteria were randomized in 1:1:1 ratio in either of the 3 arms fevipiprant 450 mg dose once daily (o.d.), fevipiprant 150 mg dose o.d. or placebo o.d. in addition to SoC (mometasone furoate spray).

The study included:

* a Screening period of 2 weeks to assess eligibility
* a Run-in period of 4 weeks where patients utilized mometasone furoate spray (200 μg once daily, administered as two 50 μg actuations into each nostril)
* a Treatment period of 16 weeks. Patients continued to use the mometasone furoate SoC throughout the treatment period.
* a Follow-up period of 2 weeks following the last dose of study drug to collect additional data for safety variables.

The purpose of this study was to evaluate the efficacy and safety of fevipiprant 150 mg and 450 mg compared to placebo in the reduction of nasal polyps size and the effect on symptoms, quality of life and smell via patient-reported outcomes in patients with nasal polyposis and concomitant asthma.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or more with a diagnosis of nasal polyps with Nasal polyp score >= 4 with minimum score of 2 in each nostril.
* Concomitant diagnosis of asthma for a period of at least 6 months prior to screening.
* Patients on stable asthma treatment of at least inhaled corticosteroids (any dose) alone for at least 6 months prior to screening or ICS for 6 months prior to screening with any required, inhaled medication (LABA, LAMA) added at least 6 weeks prior to screening.

Exclusion Criteria:

* Asthma exacerbation, within 6 weeks prior to screening, that required systemic corticosteroids, hospitalization or emergency room visit.
* Chronic/maintenance use of oral corticosteroids (OCS) defined as any continuous use of OCS for a period of 1 month or more, within 1 year of screening
* Use of biologics for asthma or any other indications, that has the potential to interfere/affect either asthma or nasal polyposis disease progression, within 6 months of screening.
* Use of medication for sino-nasal symptoms (antibiotics with or without OCS) within 30 days of screening or during the run-in period.
* Use of tetracycline or macrolide antibiotics specifically, within 8 weeks of screening.
* History of nasal surgery modifying the structure of the nose such that assessment of the nasal polyp score is not possible.
* Patients with baseline ACQ-5≥1.5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-06-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- Novartis Investigative Site, Irvine, California, United States
- Argentina (6):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Florida, Buenos Aires
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Mendoza
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Erpent
- Canada (2):
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Québec
- Czechia (3):
  - Novartis Investigative Site, Olomouc, Czech Republic
  - Novartis Investigative Site, Svitavy, Czech Republic
  - Novartis Investigative Site, Kladno
- Germany (2):
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Frankfurt
- Italy (3):
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Roma, RM
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Enschede
- Poland (2):
  - Novartis Investigative Site, Strzelce Opolskie
  - Novartis Investigative Site, Zawadzkie

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=732

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 25 investigative sites in 9 countries.
Pre-assignment Details: After the screening, participants went through a Run-in period of 4 weeks where they utilized mometasone furoate spray into each nostril. Afterwards, patients were randomized in 1:1:1 ratio in either of the 3 arms and continued to use the mometasone furoate spray.
Period: Overall Study
Arm/Group | Fevipiprant 150 mg | Fevipiprant 450 mg | Placebo
Started (All subjects who were randomized) | 32 | 34 | 32
Full Analysis Set (FAS) (All randomized subjects who received at least one dose of study treatment AND had baseline NPS score >=4) | 31 | 32 | 28
Safety Analysis Set (SAF) (All subjects who received at least one dose of study treatment) | 32 | 34 | 32
Completed | 32 | 32 | 31
Not Completed | 0 | 2 | 1
Not completed — Subject decision | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fevipiprant 150 mg | Fevipiprant 450 mg | Placebo | Total
Number analyzed (Participants) | 32 | 34 | 32 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (13.36) | 50.9 (13.10) | 48.5 (13.43) | 50.1 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 12 | 43
  Male | 16 | 19 | 20 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32 | 34 | 31 | 97
  Black | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Nasal Polyp Score at Week 16
Description: Nasal Polyp Score (NPS) is the sum of the right and left nostril scores, as evaluated by means of nasal endoscopy. Total score ranges from 0 to 8 (scored 0 [no polyp] to 4 [large polyps] for each nostril), with a lower score indicating smaller-sized polyps.
  Baseline NPS is defined as the last measurement performed on or before the date of randomization.
  A negative change from baseline in NPS is considered a favorable outcome.
Time Frame: Baseline, Week 16
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Fevipiprant 150 mg | Fevipiprant 450 mg | Placebo
Number analyzed (Participants) | 31 | 32 | 28
score on scale | 0.20 (0.224) | -0.10 (0.216) | 0.14 (0.233)
Statistical Analysis 1: Comparison: Fevipiprant 150 mg vs Placebo; Test type: Superiority; p = 0.979, Mixed Model for Repeated Measures (MMRM) — Adjusted p-value is reported. The adjusted p-value was obtained from the Dunnet Multiplicity Correction applied to control the Type I error for the primary analysis; Least Squares (LS) Mean = 0.05, 95% CI 2-sided [-0.59 to 0.70], Standard Error of Mean 0.323
Statistical Analysis 2: Comparison: Fevipiprant 450 mg vs Placebo; Test type: Superiority; p = 0.656, MMRM — [p-value comment as in outcome 1, analysis 1]; LS Mean = -0.25, 95% CI 2-sided [-0.88 to 0.39], Standard Error of Mean 0.319

2. Secondary Outcome: Change From Baseline in Nasal Congestion Score at Week 16
Description: The nasal congestion score (NCS) is assessed via a questionnaire where patients are asked "Is your nose blocked?" with responses ranging from 0 = not at all, to 3=severe.
  Baseline NCS is defined as the last assessment performed on or before the date of randomization.
  A negative change from baseline in NCS is considered a favorable outcome.
Time Frame: Baseline, Week 16
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Fevipiprant 150 mg | Fevipiprant 450 mg | Placebo
Number analyzed (Participants) | 31 | 32 | 28
score on scale | -0.15 (0.172) | -0.35 (0.171) | -0.80 (0.181)
Statistical Analysis 1: Comparison: Fevipiprant 150 mg vs Placebo; Test type: Superiority; p = 0.012, MMRM — Unadjusted p-value; LS Mean = 0.64, 95% CI 2-sided [0.15 to 1.14], Standard Error of Mean 0.249
Statistical Analysis 2: Comparison: Fevipiprant 450 mg vs Placebo; Test type: Superiority; p = 0.074, MMRM — Unadjusted p-value; LS Mean = 0.45, 95% CI 2-sided [-0.04 to 0.94], Standard Error of Mean 0.248

3. Secondary Outcome: Change From Baseline in Quality of Life as Assessed by the SNOT-22 Questionnaire at Week 16
Description: SNOT-22 (Sino-Nasal Outcome Test) Questionnaire is a disease specific Health-Related Quality of Life (HRQoL) measure that comprises a list of 22 symptoms and social or emotional consequences of the nasal disorder. Every participant is asked to rate how severe each problem had been for them over the past 2 weeks on a scale from 0 (no problem) to 5 (problem as bad as it can be). The total score is the sum of the scores for all 22 items, ranging from 0 to 110, with a lower score indicating better HRQoL.
  Baseline SNOT-22 is defined as the last assessment performed on or before the date of randomization.
  A negative change from baseline in SNOT-22 is considered a favorable outcome.
Time Frame: Baseline, Week 16
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Fevipiprant 150 mg | Fevipiprant 450 mg | Placebo
Number analyzed (Participants) | 31 | 32 | 28
score on scale | -3.23 (3.349) | -10.61 (3.358) | -8.44 (3.571)
Statistical Analysis 1: Comparison: Fevipiprant 150 mg vs Placebo; Test type: Superiority; p = 0.288, MMRM — Unadjusted p-value; LS Mean = 5.22, 95% CI 2-sided [-4.49 to 14.93], Standard Error of Mean 4.881
Statistical Analysis 2: Comparison: Fevipiprant 450 mg vs Placebo; Test type: Superiority; p = 0.661, MMRM — Unadjusted p-value; LS Mean = -2.17, 95% CI 2-sided [-11.99 to 7.65], Standard Error of Mean 4.936

4. Secondary Outcome: Change From Baseline in Sense of Smell as Assessed by the University of Pennsylvania Smell Identification Test (UPSIT) at Week 16
Description: The UPSIT (University of Pennsylvania Smell Identification Test) is a test that measures an individual's ability to detect odors. It consists of 4 workbooks of 10 pages each. On each page there is a different "scratch and sniff" strip which is embedded with a microencapsulated odorant and a question regarding the smell detected with a four-choice option for the response. The total number of questions in UPSIT is 40. The number of correct responses regarding the smells being experienced is summed to provide a total score that ranges from 0 to 40, with a higher score indicating a better sense of smell.
  Baseline UPSIT is defined as the last assessment performed on or before the date of randomization.
  A positive change from baseline in UPSIT is considered a favorable outcome.
Time Frame: Baseline, Week 16
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on scale
Arm/Group | Fevipiprant 150 mg | Fevipiprant 450 mg | Placebo
Number analyzed (Participants) | 31 | 32 | 28
score on scale | 1.05 (1.242) | 4.95 (1.259) | 0.44 (1.315)
Statistical Analysis 1: Comparison: Fevipiprant 150 mg vs Placebo; Test type: Superiority; p = 0.735, MMRM — Unadjusted p-value; LS Mean = 0.61, 95% CI 2-sided [-2.98 to 4.21], Standard Error of Mean 1.809
Statistical Analysis 2: Comparison: Fevipiprant 450 mg vs Placebo; Test type: Superiority; p = 0.015, MMRM — Unadjusted p-value; LS Mean = 4.51, 95% CI 2-sided [0.89 to 8.13], Standard Error of Mean 1.821

ADVERSE EVENTS:
Time Frame: From first dose of study treatment until end of study treatment plus 2 weeks post treatment, up to Week 18.
Description: Any sign or symptom that occurs during the study treatment plus 2 weeks post treatment.
Arm/Group | Fevipiprant 150 mg | Fevipiprant 450 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34 | 0/32
Other Adverse Events (participants affected / at risk) | 17/32 | 13/34 | 11/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fevipiprant 150 mg (N=32) | Fevipiprant 450 mg (N=34) | Placebo (N=32)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Tongue discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Gastric infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 2
Laryngitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2
Oral herpes (Infections and infestations) | 1 | 2 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 2
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Amylase increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 0
Weight increased (Investigations) | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT03681093/Prot_001.pdf
  • Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT03681093/SAP_000.pdf